CLINICAL TRIAL: NCT01204814
Title: Prevalence of HIV-1 Drug Resistance Within a Female Screening Population for HIV Prevention Trials
Brief Title: HIV-1 Resistance at Screening for HIV Prevention Studies
Status: Completed | Type: Observational
Sponsor: Microbicide Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: MTN-009; 5U01AI068633-04 (NIH)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: HIV
Keywords: HIV; Drug resistance; mutations; ARV's

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood Plasma
Oversight: Data Monitoring Committee: Yes

SUMMARY:
MTN-009 is a multi-site, cross-sectional study that will provide an estimate of the prevalence of ARV resistance in the population of women who present to study sites to be pre-screened or screened for participation in an HIV prevention trial. To date, a comprehensive surveillance of HIV drug resistance in newly diagnosed women of reproductive age has yet to be undertaken. The primary goal of MTN-009 is to assess the frequency of HIV drug resistance mutations among women who test HIV-positive when presenting to screen for participation in HIV prevention trials.

DETAILED DESCRIPTION:
MTN-009 is a multi-site, cross-sectional study that will provide an estimate of the prevalence of ARV resistance in the population of women who present to study sites to be pre-screened or screened for participation in an HIV prevention trial. To date, a comprehensive surveillance of HIV drug resistance in newly diagnosed women of reproductive age has yet to be undertaken. The primary goal of MTN-009 is to assess the frequency of HIV drug resistance mutations among women who test HIV-positive when presenting to screen for participation in HIV prevention trials. Secondary aims include the identification and evaluation of behavioral indicators including self or sexual partner(s) exposures to antiretroviral (ARV) drugs as risk factors for drug resistant HIV infection, as well as the characterization of the degree of immunodeficiency and risk of disease progression by quantifying plasma HIV-1 RNA and CD4-positive T cells among women who test HIV-positive when presenting to screen for participation in an HIV prevention trial. Exploratory aims include the identification of polymorphic or subtype-specific sequence changes in HIV-1 that may impact susceptibility to ARVs, and the estimation of the proportion of HIV-positive women who have chronic versus recent HIV infection.

The finding of significant resistance, or lack thereof, to ARV-based study products delivered vaginally or taken orally may guide decisions related to future microbicide and PrEP studies. In addition, MTN-009 will provide valuable comparison data for the resistance data obtained in MTN-015, the MTN seroconverter study.

ELIGIBILITY:
Inclusion Criteria:

* Present to an MTN-009 study site to pre-screen or screen for an HIV prevention trial
* Age 18-40 years, verified per site standard operating procedures (SOP)
* Able and willing to provide written informed consent for participation in MTN-009
* Able and willing to provide adequate locator information, as defined in site SOPs

Exclusion Criteria:

* Any condition that, in the investigator's opinion, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achievement of the study objectives

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women of reproductive age who are interested in participating in HIV prevention trials
Sampling Method: Non-Probability Sample
Enrollment: 1074 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To assess the frequency of HIV drug resistance mutations among women who test HIV-positive when presenting to screen for participation in HIV prevention trials | 2 years
  Mutations in HIV-1 reverse transcriptase and protease known to be associated with drug resistance

SECONDARY OUTCOMES:
To identify and evaluate behavioral indicators including self or sexual partner(s) exposures to ARV drugs as risk factors for drug resistant HIV infection in women who present for screening to participate in HIV prevention trials | 2 years
  Participant self-reported ARV drug exposures and other behaviors or herself or sexual partner(s) that may be associated with risk of drug resistant HIV-1 infections
• To characterize the degree of immunodeficiency and risk of disease progression by quantifying plasma HIV-1 RNA and CD4-positive T cells among women who test HIV-positive when presenting for screening to participate in HIV prevention trials | 2 years
  • Plasma HIV-1 RNA levels and CD4-positive T cell counts
  Plasma HIV-1 RNA levels and CD4-positive T cell counts

CONTACTS AND LOCATIONS:
Overall Officials: Urvi Parikh, PhD, Study Chair — MTN Virology CORE
Locations (7):
- South Africa (7):
  - South African Medical Research Council, HIV Prevention Research Unit, Durban, KwaZulu-Natal
  - South African Medical Research Council, Botha's Hill, Durban, KwaZulu-Natal
  - South African Medical Research Council, Isipingo, Durban, KwaZulu-Natal
  - South African Medical Research Council, RK Khan (Chatsworth), Durban, KwaZulu-Natal
  - South African Medical Research Council, Umkomaas, Durban, KwaZulu-Natal
  - South African Medical Research Council, Verulam, Durban, KwaZulu-Natal
  - South African Medical Research Council, Tongaat, KwaZulu-Natal

REFERENCES:
- [Result] Parikh UM, Kiepiela P, Ganesh S, Gomez K, Horn S, Eskay K, Kelly C, Mensch B, Gorbach P, Soto-Torres L, Ramjee G, Mellors JW; MTN-009 Protocol Team. Prevalence of HIV-1 drug resistance among women screening for HIV prevention trials in KwaZulu-Natal, South Africa (MTN-009). PLoS One. 2013 Apr 9;8(4):e59787. doi: 10.1371/journal.pone.0059787. Print 2013. PMID 23585827
- [Result] Mensch BS, Gorbach PM, Kelly C, Kiepiela P, Gomez K, Ramjee G, Ganesh S, Morar N, Soto-Torres L, Parikh UM. Characteristics Associated with HIV Drug Resistance Among Women Screening for an HIV Prevention Trial in KwaZulu-Natal, South Africa. AIDS Behav. 2015 Nov;19(11):2076-86. doi: 10.1007/s10461-015-1056-4. PMID 25931240